CLINICAL TRIAL: NCT00322101
Title: A Multi-center Phase III Study Comparing Myeloablative to Nonmyeloablative Transplant Conditioning in Patients With Myelodysplastic Syndrome or Acute Myelogenous Leukemia
Brief Title: Low-Dose or High-Dose Conditioning Followed by Peripheral Blood Stem Cell Transplant in Treating Patients With Myelodysplastic Syndrome or Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1992.00; NCI-2010-00737 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01CA078902 (NIH); K23HL084054 (NIH); P01CA018029 (NIH); P01HL036444 (NIH)
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2013-10-28 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Acute Myeloid Leukemia/Transient Myeloproliferative Disorder; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Childhood Acute Myeloid Leukemia in Remission; Childhood Myelodysplastic Syndromes; de Novo Myelodysplastic Syndromes; Myelodysplastic Syndrome With Isolated Del(5q); Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myeloproliferative Syndrome, Transient; Congenital Abnormalities; Chromosome 5q Deletion Syndrome; Myeloproliferative Disorders | interventions — Whole-Body Irradiation; Cyclophosphamide; Mycophenolic Acid; Busulfan; Cyclosporine; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation; Cytogenetic Analysis; Flow Cytometry; In Situ Hybridization, Fluorescence; Amplified Fragment Length Polymorphism Analysis; Tacrolimus; Methotrexate; merphos

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Nonmyeloablative regimen) (Experimental): CONDITIONING: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo low-dose total-body irradiation on day 0.
  TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell (PBSC) infusion on day 0.
  GRAFT-VS-HOST DISEASE PROPHYLAXIS: Patients receive cyclosporine every 12 hours on days -3 to 57 with taper on days 57-177 or cyclosporine every 12 hours on days -3 to 100 with taper on days 101-177. Patients also receive oral mycophenolate mofetil every 12 hours on days 0-27 or every 8 hours on days 0-40 with taper on days 41-96.
  Interventions: Radiation: total-body irradiation; Drug: mycophenolate mofetil; Drug: cyclosporine; Drug: fludarabine phosphate; Procedure: peripheral blood stem cell transplantation; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Other: laboratory biomarker analysis; Genetic: cytogenetic analysis; Other: flow cytometry; Genetic: fluorescence in situ hybridization; Other: pharmacological study; Genetic: polymorphism analysis
- Arm II (Myeloablative regimen) (Experimental): CONDITIONING: Patients are assigned to 1 of 2 treatment groups.
  Group A: Patients receive fludarabine IV once daily and oral busulfan four times daily or busulfan IV over 3 hours on days -5 to -2.
  Group B: Patients receive cyclophosphamide IV over 1-2 hours on days -3 and -2 and oral busulfan four times daily or busulfan IV over 3 hours on days -7 to -4.
  TRANSPLANTATION: Patients undergo PBSC infusion on day 0.
  GRAFT-VS-HOST DISEASE PROPHYLAXIS: Patients receive tacrolimus IV continuously or orally every 12 hours on days -1 to 56 and taper on days 57-200. Patients also receive methotrexate IV on days 1, 3, 6, and 11.
  Interventions: Procedure: allogeneic hematopoietic stem cell transplantation; Drug: cyclophosphamide; Drug: busulfan; Drug: fludarabine phosphate; Procedure: peripheral blood stem cell transplantation; Other: laboratory biomarker analysis; Other: flow cytometry; Genetic: fluorescence in situ hybridization; Other: pharmacological study; Genetic: polymorphism analysis; Drug: tacrolimus; Drug: methotrexate

INTERVENTIONS:
Radiation: total-body irradiation — Radiation
  Other Names: TBI
  Arms: Arm I (Nonmyeloablative regimen)
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic transplantation
  Arms: Arm II (Myeloablative regimen)
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
  Arms: Arm II (Myeloablative regimen)
Drug: mycophenolate mofetil — Given orally
  Other Names: Cellcept; MMF
  Arms: Arm I (Nonmyeloablative regimen)
Drug: busulfan — Given IV or orally
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
  Arms: Arm II (Myeloablative regimen)
Drug: cyclosporine — Given IV or orally
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
  Arms: Arm I (Nonmyeloablative regimen)
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Procedure: peripheral blood stem cell transplantation — Undergo transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — Undergo allogeneic transplantation
  Arms: Arm I (Nonmyeloablative regimen)
Other: laboratory biomarker analysis — Correlative studies
Genetic: cytogenetic analysis — Correlative studies
  Arms: Arm I (Nonmyeloablative regimen)
Other: flow cytometry — Correlative studies
Genetic: fluorescence in situ hybridization — Correlative studies
  Other Names: fluorescence in situ hybridization (FISH)
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Genetic: polymorphism analysis — Correlative studies
Drug: tacrolimus — Given IV or orally
  Other Names: FK 506; Prograf
  Arms: Arm II (Myeloablative regimen)
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
  Arms: Arm II (Myeloablative regimen)

SUMMARY:
RATIONALE: Giving chemotherapy, such as fludarabine phosphate, busulfan, and cyclophosphamide, and total-body radiation therapy before a donor peripheral stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. It is not yet known whether low-dose chemotherapy and total-body radiation therapy is more effective than high-dose chemotherapy in treating patients with myelodysplastic syndrome or acute myeloid leukemia.

PURPOSE: This phase III trial is studying low-dose conditioning to see how well it works compared to high-dose conditioning followed by peripheral blood stem cell transplant in treating patients with myelodysplastic syndromes or acute myeloid leukemia

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine whether the conditioning intensity affects outcomes after HCT in patients with MDS or AML who have < 5% marrow myeloblasts at the time of HCT.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

Arm I (Nonmyeloablative regimen):

CONDITIONING: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo low-dose total-body irradiation on day 0.

TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell (PBSC) infusion on day 0.

GRAFT-VS-HOST DISEASE PROPHYLAXIS: Patients receive cyclosporine every 12 hours on days -3 to 57 with taper on days 57-177 or cyclosporine every 12 hours on days -3 to 100 with taper on days 101-177. Patients also receive oral mycophenolate mofetil every 12 hours on days 0-27 or every 8 hours on days 0-40 with taper on days 41-96.

Arm II (Myeloablative regimen):

CONDITIONING: Patients are assigned to 1 of 2 treatment groups.

Group A: Patients receive fludarabine IV once daily and oral busulfan four times daily or busulfan IV over 3 hours on days -5 to -2.

Group B: Patients receive cyclophosphamide IV over 1-2 hours on days -3 and -2 and oral busulfan four times daily or busulfan IV over 3 hours on days -7 to -4.

TRANSPLANTATION: Patients undergo PBSC infusion on day 0.

GRAFT-VS-HOST DISEASE PROPHYLAXIS: Patients receive tacrolimus IV continuously or orally every 12 hours on days -1 to 56 and taper on days 57-200. Patients also receive methotrexate IV on days 1, 3, 6, and 11.

Treatment in both arms continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Myelodysplastic syndrome (MDS) or transformed acute myelogenous leukemia (transformed from MDS)
* De novo acute myelogenous leukemia (AML) beyond first remission
* Intermediate or high risk de novo AML in first complete response (at FHCRC unrelated donor recipients only)
* Chemotherapy required prior to HCT for all patients:
* A) Interval between start of a cycle of cytoreductive chemotherapy and infusion of donor stem cells must be at least 30 days; chemotherapy received for disease maintenance will be allowed during this time period
* B) All patients must have < 5% myeloblasts based on marrow morphology performed within 21 days prior to start of conditioning regimen and at least 3-4 weeks after the start of pre-transplant cytoreductive chemotherapy
* C) All patients must have no circulating peripheral blood myeloblasts present based on morphologic analysis
* Age 65 years or under for patients with related donors; age 60 years or under for patients with unrelated donors
* HCT-Specific Comorbidity Index Score (HCT-CI) < 3
* Related donor (age > 12 years, nonsyngeneic) or unrelated donor, HLA phenotypically or genotypically identical at the allele level at A,B,C,DRQ1, and CBQ1
* DONOR: Related or unrelated donors who are genotypically or phenotypically matched by high resolution HLA typing (HLA-A, B, C, DRB1, and DQB1); class 1 single allele mismatch allowed
* DONOR: Patient and donor pairs homozygous at a mismatched allele in the graft rejection vector are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0201, and this type of mismatch is not allowed
* DONOR: A positive anti-donor cytotoxic crossmatch or flow cytometric assay is an absolute donor exclusion at FHCRC/SCCA
* DONOR: Age >= 12 years
* DONOR: Donors must consent to PBSC mobilization with G-CSF and leukaphereses; bone marrow as a source of stem cells will not be allowed
* DONOR: Donor must have adequate veins for leukaphereses or agree to placement of central venous catheter (femoral, subclavian)

Exclusion Criteria:

* HIV seropositivity
* Fungal infections with radiographic progression after appropriate therapy for greater than one month
* Organ dysfunction
* Symptomatic coronary artery disease or ejection fraction < 35%
* DLCO < 65%, FEV1 < 65% or receiving supplementary continuous oxygen
* Liver function abnormalities: Patients with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, histology, and the degree of portal hypertension; patients with fulminant liver failure, cirrhosis with evidence of portal hypertension or bridging fibrosis, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, and symptomatic biliary disease will be excluded
* Karnofsky Performance Score < 70
* Lansky-Play Performance Score < 70 for pediatric patients
* Life expectancy severely limited (< 2 years) by disease other than MDS/AML
* Fertile men and women unwilling to use contraceptive techniques during and for 12 months following treatment
* Patients with active non-hematological malignancies except:
* A) Patients with follicular or low grade lymphoma will be eligible as long as they have not and do not require active treatment for control of their disease
* B) Patients with localized non-melanoma skin malignancies
* Patients with poorly controlled hypertension who are unable to have blood pressure stabilized below 150/90 mm Hg on standard medication
* Females who are pregnant or breastfeeding
* Patients with systemic, uncontrolled infections
* Active CNS disease as identified by positive CSF cytospin
* DONOR: Identical twin
* DONOR: Age < 12 years
* DONOR: Pregnancy
* DONOR: HIV seropositivity
* DONOR: Inability to achieve adequate venous access
* DONOR: Known adverse reaction to G-CSF

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-01; Primary Completion 2012-04 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Scott, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (8):
- United States (7):
  - HealthOne Presbyterian St. Lukes Medical Center, Denver, Colorado
  - Emory University, Altanta, Georgia
  - Weill Cornell University, New York, New York
  - University of Utah, Salt Lake City, Utah
  - Veterans Administration Center-Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Medical College Wisconsin, Milwaukee, Wisconsin
- Technical University Dresden, Dresden, Saxony, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from medical clinics while being evaluated for stem cell transplantation
Period: Overall Study
Arm/Group | Arm I (Nonmyeloablative Regimen) | Arm II (Myeloablative Regimen)
Started | 14 | 11
Completed | 14 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Nonmyeloablative Regimen) | Arm II (Myeloablative Regimen) | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.47 (9.49) | 52.82 (5.78) | 52.2 (7.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15
  Germany | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: At 2 years
Population: 2 patients in the nonmyeloablative arm did not receive transplant due to relapse and withdrawal of consent
Measure: Number; unit: participants
Arm/Group | Arm I (Nonmyeloablative Regimen) | Arm II (Myeloablative Regimen)
Number analyzed (Participants) | 12 | 11
participants | 6 | 6

2. Secondary Outcome: Progression-free Survival
Description: IWG criteria was used to determine disease progression
Time Frame: After stem cell infusion to date of last follow up.
Population: 2 patients in the nonmyeloablative arm did not receive a transplant due to relapse and withdrawal of consent
Measure: Number; unit: participants
Arm/Group | Arm I (Nonmyeloablative Regimen) | Arm II (Myeloablative Regimen)
Number analyzed (Participants) | 12 | 11
participants | 7 | 5

3. Secondary Outcome: Non-relapse Mortality
Time Frame: At 100 days
Population: 2 patients in the nonmyeloablative arm did not receive transplant due to relapse and withdrawal of consent
Measure: Number; unit: participants
Arm/Group | Arm I (Nonmyeloablative Regimen) | Arm II (Myeloablative Regimen)
Number analyzed (Participants) | 12 | 11
participants | 0 | 0

4. Secondary Outcome: Donor Cell Engraftment
Description: Chimerism analysis was performed in patients who recieved nonmyeloablative tranplsnat. In this group the definition of engraftment was a CD3 count greater than 50%. In the myeloablative group, engraftment was defined as an absolute neutrophil count greater than 50%.
Time Frame: After stem cell infusion to day 28
Population: 2 patients who were randomized to receive nonmyeloablative conditioning did not undergo transplant due to relapse and withdrawal of consent
Measure: Number; unit: participants
Arm/Group | Arm I (Nonmyeloablative Regimen) | Arm II (Myeloablative Regimen)
Number analyzed (Participants) | 12 | 11
participants | 11 | 11

5. Secondary Outcome: Incidence of Disease Progression/Relapse
Description: Disease progression/relapse was defined by IWG criteria
Time Frame: After stem cell infusion to date of last follow up.
Measure: Number; unit: participants
Arm/Group | Arm I (Nonmyeloablative Regimen) | Arm II (Myeloablative Regimen)
Number analyzed (Participants) | 12 | 11
participants | 7 | 2

6. Secondary Outcome: Incidence and Severity of Acute and Chronic Graft-vs-host Disease
Time Frame: After transplantation
Measure: Number; unit: participants
Arm/Group | Arm I (Nonmyeloablative Regimen) | Arm II (Myeloablative Regimen)
Number analyzed (Participants) | 12 | 11
participants | 1 | 4

ADVERSE EVENTS:
Arm/Group | Arm I (Nonmyeloablative Regimen) | Arm II (Myeloablative Regimen)
Serious Adverse Events (participants affected / at risk) | 3/12 | 4/11
Other Adverse Events (participants affected / at risk) | 12/12 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Nonmyeloablative Regimen) (N=12) | Arm II (Myeloablative Regimen) (N=11)
severe diarrhea due to gut GVHD (Gastrointestinal disorders) | 2 (2) | 2 (2)
tachycardia and hypotenstion (Cardiac disorders) | 1 (1) | 0 (0)
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Nonmyeloablative Regimen) (N=12) | Arm II (Myeloablative Regimen) (N=11)
Mucositis (Gastrointestinal disorders) | 0 (0) | 6 (6)
Infection (Infections and infestations) | 12 (12) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes